CLINICAL TRIAL: NCT04844957
Title: Correlation Between Vitamin D and Symptoms Severity of Autonomic Nervous Mediated Syncope（NMS） Child and it 's RAAS
Brief Title: Correlation Between Vitamin D and Symptoms Severity of Autonomic Nervous Mediated Syncope Child and it 's RAAS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kongyujie (Other)
Collaborators: LanZhou University (Other)
Responsible Party: Sponsor-Investigator, Kongyujie, Graduate student, LanZhou University
Organization: LanZhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021A-057
Record Dates: First submitted 2021-03-28; First posted 2021-04-14 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Vitamin D
Keywords: children ; VVS； vitamin D ; symptom score ; RAAS
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Clinical Study of Vitamin D in Children With NMS (Other): Correlation between vitamin D and symptoms severity of autonomic nervous mediated syncope child and it 's RAAS
  Interventions: Drug: Vitamin D; Device: Full automatic chemiluminescence measuring instrument

INTERVENTIONS:
Drug: Vitamin D — Clinical Study
  Other Names: Vitamin D drops
Device: Full automatic chemiluminescence measuring instrument — Chemiluminescence immunoassay

SUMMARY:
children ; autonomic nervous mediated syncope； vitamin D ; symptom score ; renin-angiotensin-aldosterone-system

DETAILED DESCRIPTION:
children with autonomic nervous mediated syncope have seriously affects children's physical and mental health and quality of life, and the incidence rate is also increasing year by year. But the current treatment measures are not ideal, Therefore, we need to look for new biological indicators, according to different biological indicators to develop different treatment options, so as to improve the current situation of poor treatment of children with NMS

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with OI;
* Compliance with the diagnostic guidelines for Syncope in children (2016 edition) and 2018 syncope in children and adolescents in the cardiovascular group of the Society of Pediatrics, Chinese Medical Association The diagnostic criteria of Oi in the Diagnostic and therapeutic guidelines.

Exclusion Criteria:

* Taken 3 months prior to admission Vitamin D or hormone drugs;
* Heart, brain, nerves, metabolism, blood and other apparatus Syncope or aura of syncope caused by a qualitative disease;

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Vitamin D levels | 3 months after taking the drug
  Vitamin D levels after supplementation

SECONDARY OUTCOMES:
RAAS levels | 3 months after taking the drug
  RAAS levels after vitamin D supplementation

OTHER OUTCOMES:
OI symptom scores | 3 months after taking the drug
  OI symptom scores after vitamin D supplementation

CONTACTS AND LOCATIONS:
Overall Officials: xiangyu Dong, Professor, Study Director — LanZhou University
Locations (1):
- Kongyujie, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
Experimental outcomes